CLINICAL TRIAL: NCT01559311
Title: Efficacy of the Presence of Right Ventricular Apical Pacing Induced Ventricular Dyssynchrony as a Guiding Parameter for Biventricular Pacing in Patients With Bradycardia and Normal Ejection Fraction
Brief Title: ENHANCE-Efficacy of the Presence of Right Ventricular Apical Pacing Induced Ventricular Dyssynchrony as a Guiding Parameter for Biventricular Pacing in Patients With Bradycardia and Normal Ejection Fraction
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CR-10-003-AP-HF
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Bradycardia
Keywords: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRT-P OFF (Active Comparator): Patients randomized into the Echo-guided Group were implanted with a CRT-P device (St. Jude Medical), which was programmed to DDDR pacing mode (CRT-P OFF) at implant. For each Echo-guided Group patient, presence of RVA pacing induced ventricular dyssynchrony was assessed within 24-hour of implant using the standardized criteria of Doppler echocardiography. The Echocardiography Core Laboratory (Echo Core Lab) then analyzed each image and the treatment allocation of the Echo-guided Group was done within 72-hour post implant based on the Echo Core Lab outcomes:
  • Patients with the absence of RVA pacing induced ventricular dyssynchrony were allocated to the DDDR standard therapy with CRT-P remained OFF
  Interventions: Device: CRT-P OFF
- CRT-P ON (Experimental): Patients randomized into the Echo-guided Group were implanted with a CRT-P device (St. Jude Medical), which was programmed to DDDR pacing mode (CRT-P OFF) at implant. For each Echo-guided Group patient, presence of RVA pacing induced ventricular dyssynchrony was assessed within 24-hour of implant using the standardized criteria of Doppler echocardiography. The Echocardiography Core Laboratory (Echo Core Lab) then analyzed each image and the treatment allocation of the Echo-guided Group was done within 72-hour post implant based on the Echo Core Lab outcomes:
  • Patients with the presence of RVA pacing induced ventricular dyssynchrony were allocated to the CRT-P standard therapy with CRT-P turned ON
  Interventions: Device: CRT-P ON
- DDDR (Active Comparator): Patients randomized into the Control Group were implanted with a DDDR device (St. Jude Medical) standard therapy.
  Interventions: Device: DDDR

INTERVENTIONS:
Device: CRT-P OFF — CRT Pacemaker
  Arms: CRT-P OFF
Device: CRT-P ON — CRT Pacemaker
  Arms: CRT-P ON
Device: DDDR — Dual-chamber, rate-modulated pacemaker
  Arms: DDDR

SUMMARY:
The purpose of this clinical project is to evaluate the efficacy of the presence of Right Ventricular Apical (RVA) pacing induced ventricular dyssynchrony as a guiding parameter for bi-ventricular pacing in patients with bradycardia and normal left ventricular ejection fraction (LVEF). The results of this project may provide with the evidence based medicine for guidelines expansion of using Cardiac resynchronization therapy (CRT) in patients with Heart Block and normal LVEF (LVEF >45%).

DETAILED DESCRIPTION:
All eligible patients willing to provide written informed consent were invited to participate in the study, and then randomized 1:2 to either the Control Group or Echo-guided Group. Patients randomized into the Control Group were implanted with a dual chamber pacemaker (DDDR) device (St. Jude Medical) standard therapy. Patients randomized into the Echo-guided Group were implanted with a cardiac resynchronization therapy pacemaker (CRT-P) device (St. Jude Medical), which was programmed to DDDR pacing mode (CRT-P OFF) at implant. For each Echo-guided Group patient, presence of RVA pacing induced ventricular dyssynchrony was assessed within 24-hour of implant using the standardized criteria of Doppler echocardiography. The Echocardiography Core Laboratory (Echo Core Lab) then analyzed each image and the treatment allocation of the Echo-guided Group was done within 72-hour post implant based on the Echo Core Lab outcomes:

* Patients with the presence of RVA pacing induced ventricular dyssynchrony were allocated to the CRT-P standard therapy with CRT-P turned ON
* Patients with the absence of RVA pacing induced ventricular dyssynchrony were allocated to the DDDR standard therapy with CRT-P remained OFF

Patients meeting all the inclusion criteria and not meeting any of the exclusion criteria were eligible for the study. Data was collected at the following study visits:Enrollment, Implant & Randomization, Pre-discharge (PDH) (≤ 72 hours post implant), Month 1 follow-up visit: 30 ± 14 days post implant, Month 3 follow-up visit: 90 ± 14 days post implant, Month 6 follow-up visit: 180 ± 14 days post implant and Month 12 follow-up visit: 365 ± 14 days post implant

ELIGIBILITY:
Inclusion Criteria:

* Patient meets current indications for implantation of a DDDR pacemaker
* Patient is geographically stable and willing to comply with the required follow-up schedule
* Patient has LVEF >45%
* Patient has atrioventricular block (IIo or above)
* Patient has adequate echocardiographic images to measure LV volumes and LVEF

Exclusion Criteria:

* Patient has permanent atrial fibrillation (AF)
* Patient has unstable angina or an acute coronary syndrome
* Patient has undergone percutaneous coronary intervention or coronary artery bypass surgery within the previous 3 months
* Patient's life expectancy is less than 1 year
* Patient is less than 18 years old
* Patient is pregnant
* Patient has received a heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Man Yu, MD, Principal Investigator — Department of Medicine and Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, New Territories, Hong Kong
Locations (7):
- The Prince Charles Hospital, Chermside, Australia
- Prince of Wales Hospital, Hong Kong, China
- India (3):
  - Madras Medical Mission, Chennai
  - CARE Banjara, Hyderabad
  - All India Institute of Medical Sciences, New Delhi
- Istituto Clinico Humanitas, Rozzano, Italy
- Siriraj Hospital, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment target was 177 patients. There were 8 centers from Asia Pacific and 1 center from Italy in the study. From Feb 2013 to Dec 2014, only 98 subjects out of 177 target enrolments were recruited into the study. Sample size was not reached due to difficulty in enrollment.
Groups:
- CRT-P OFF: Echo-guided Group - Dual chamber pacemaker (DDDR) Standard Therapy
- CRT-P ON: Echo-guided Group - Cardiac resynchronization therapy pacemaker (CRT-P) Standard Therapy
- DDDR: Control Group - DDDR Standard Therapy
Period: Overall Study
Arm/Group | CRT-P OFF | CRT-P ON | DDDR
Started | 30 (Enrollment & Baseline) | 34 (Enrollment & Baseline) | 34 (Enrollment & Baseline)
Implant | 28 | 34 | 32
1-Month | 27 | 34 | 29
3-Month | 27 | 34 | 29
6-Month | 27 | 33 | 28
Completed | 27 (12-Month) | 28 (12-Month) | 26 (12-Month)
Not Completed | 3 | 6 | 8
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Difficulty in cannulating the lateral ve | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Death | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Age = (the year of visit - year of birth)
Groups:
- CRT-P OFF: Echo-guided Group - DDDR Standard Therapy
- CRT-P ON: Echo-guided Group - CRT-P Standard Therapy
- Total: Total of all reporting groups
Arm/Group | CRT-P OFF | CRT-P ON | DDDR | Total
Number analyzed (Participants) | 30 | 34 | 34 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.53 (11.99) | 68.41 (13.22) | 72.29 (9.84) | 69.49 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 12 | 36
  Male | 20 | 20 | 22 | 62
Atrial Fibrillation History [Number; unit: participants]
  None | 30 | 32 | 33 | 95
  Paroxysmal | 0 | 2 | 1 | 3
Heart Rate [Mean (Standard Deviation); unit: bpm] | 47.37 (16.55) | 47.68 (10.35) | 49 (14.64) | 48.04 (13.85)
Rhythm on 12-lead ECG [Number; unit: participants]
  Sinus | 7 | 11 | 10 | 28
  Atrial Fibrillation | 0 | 0 | 1 | 1
  2:1 Heart Block | 5 | 4 | 6 | 15
  2nd Degree Heart Block | 3 | 2 | 1 | 6
  Complete Heart Block | 11 | 14 | 12 | 37
  Atrioventricular Dissociation (AVD) | 0 | 0 | 1 | 1
  Intermitent Pacing | 0 | 0 | 1 | 1
  Complete Heart Block with Escape Rhythm | 1 | 0 | 0 | 1
  Complete AV block with junctional escape | 0 | 1 | 0 | 1
  Ventricular Paced rhythm | 0 | 1 | 0 | 1
  Sinus Bradycardia | 1 | 0 | 1 | 2
  Wenkebach | 2 | 0 | 1 | 3
  Heart Block | 0 | 1 | 0 | 1
PR interval [Mean (Standard Deviation); unit: ms] — Population: The population for this measure differs from overall number of baseline participants because of missing data
  ms
    number analyzed (Participants) | 15 | 22 | 17 | 54
    (all) | 227.60 (78.50) | 236.27 (80.99) | 214.76 (56.42) | 227.09 (72.60)
QRS interval [Mean (Standard Deviation); unit: ms] | 114.67 (29.83) | 118.82 (40.06) | 131.47 (36.56) | 121.94 (36.31)
Baseline Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 65.19 (8.42) | 63.14 (8.70) | 64.72 (7.51) | 64.31 (8.18)
Baseline Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: ml] | 32.93 (15.92) | 41.55 (20.22) | 36.92 (23.85) | 37.31 (20.51)
Baseline Left Ventricular End Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: ml] | 84.72 (31.14) | 104.28 (34.08) | 88.78 (35.27) | 92.91 (34.36)

OUTCOME MEASURES:

1. Primary Outcome: LVEF
Description: Left Ventricular Ejection Fraction (LVEF) for assessment of Left ventricular (LV) systolic function
Time Frame: 12 months
Population: From Feb 2013 to Dec 2014, only 98 subjects out of 177 target enrolments were recruited into the study.
Measure: Mean (Standard Deviation); unit: % LVEF
Arm/Group | CRT-P OFF | CRT-P ON | DDDR
Number analyzed (Participants) | 27 | 28 | 26
% LVEF | 64.22 (7.53) | 63.14 (7.51) | 59.96 (10.47)
Statistical Analysis 1: Comparison: CRT-P ON vs DDDR; * H01: μ LVEF, 1= μ LVEF, 2a vs H1a: μ LVEF, 1 < μ LVEF, 2a * Where μ LVEF, 1 is the mean of LVEF at month 12 in DDDR Gp. * μ LVEF, 2a is the mean of LVEF at month 12 in CRT-P ON Gp,; Test type: Superiority or Other; p = 0.1734, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CRT-P OFF vs DDDR; * H03: μ LVEF, 1= μ LVEF, 2b vs H1a: μ LVEF, 1 < μ LVEF, 2b * Where μ LVEF, 1 is the mean of LVEF at month 12 in DDDR Gp. * μ LVEF, 2b is the mean of LVEF at month 12 in the CRT-P OFF Gp; Test type: Superiority or Other; p = 0.1439, Wilcoxon (Mann-Whitney)

2. Primary Outcome: LVESV
Description: Left ventricular end-systolic volume (LVESV) for assessment of LV remodeling
Time Frame: 12 months
Population: From Feb 2013 to Dec 2014, only 98 subjects out of 177 target enrolments were recruited into the study.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | CRT-P OFF | CRT-P ON | DDDR
Number analyzed (Participants) | 27 | 28 | 26
ml | 30.52 (14.73) | 34.54 (14.74) | 36.38 (21.73)
Statistical Analysis 1: Comparison: CRT-P ON vs DDDR; * H02: μ LVESV, 1 = μ LVESV, 2a vs H1b: μ LVESV, 1 > μ LVESV, 2a * Where, μLVESV, 1 is the mean of LVESV at month 12 in the DDDR Group, * μLVESV, 2a is the mean of LVESV at month 12 in the CRT-P ON group; Test type: Superiority or Other; p = 0.6276, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CRT-P OFF vs DDDR; * H04: μ LVESV, 1 = μ LVESV, 2b vs H1b: μ LVESV, 1 > μ LVESV, 2b * Where, μLVESV, 1 is the mean of LVESV at month 12 in the DDDR Group, * and μLVESV, 2b is the mean of LVESV at month 12 in CRT-P OFF group; Test type: Superiority or Other; p = 0.5871, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 Months Follow Up
Arm/Group | CRT-P OFF | CRT-P ON | DDDR
Serious Adverse Events (participants affected / at risk) | 5/30 | 11/34 | 12/34
Other Adverse Events (participants affected / at risk) | 10/30 | 18/34 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-P OFF (N=30) | CRT-P ON (N=34) | DDDR (N=34)
Acute renal failure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atypical chest pain (General disorders) | 1 (6) | 0 (0) | 1 (1)
Coronary Artery Disease (CAD) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diaphragmatic/ phrenic stimulation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extrusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatty liver (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hematoma (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypervolemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 1 (2)
Infected osteoradionecrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Knee effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lead dislodgement (General disorders) | 0 (0) | 2 (2) | 2 (2)
Lead repositioning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non ST-segment elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Renal imairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Supraglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-P OFF (N=30) | CRT-P ON (N=34) | DDDR (N=34)
Abnormal liver function tests (LFTs) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Accidental injury (General disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronary sinus dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased LVEF (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Degenerative myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic/ phrenic stimulation (General disorders) | 0 (0) | 2 (3) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Elbow and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Enlarged prostate (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye itching (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Frozen sholder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Globus sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glucosuria (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hematoma (General disorders) | 1 (1) | 3 (3) | 1 (1)
Hemorrhoid (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lead dislodgement (General disorders) | 1 (1) | 1 (1) | 1 (1)
Lead fixation difficulty (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medication induced side effects (General disorders) | 1 (2) | 1 (1) | 0 (0)
Metabolic acidosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mode switch (General disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peri-rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Suspected cancer (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 0 (0) | 1 (1)
Threshold increase (General disorders) | 0 (0) | 3 (3) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Varicella Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle cramps (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size was not reached due to difficulty in enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less